CLINICAL TRIAL: NCT04134455
Title: The Mesh-RTL Project for Prevention of Incisional Hernia: Clinical Trial of Non-inferiority to Compare Two Aponeurotic Closure Techniques in Midline Laparotomy in Patients With Elevated Risk for Hernia
Brief Title: The Mesh-RTL Project, for Prevention of Incisional Hernia
Acronym: RTL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Principal Investigator, Edgard Lozada, Master in clinical research, Hospital Regional de Alta Especialidad del Bajio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI/HRAEB/2018/08; MeshVsRTL (Other: Hraeb)
Record Dates: First submitted 2019-10-08; First posted 2019-10-22 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Hernia Incisional
Keywords: Mesh; RTL(reinforced tension line); Prevention; Prophylactic Mesh
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Intervention Model Description: Clinical trial of non-inferiority
Who Masked: Participant, Investigator
Masking Description: The participant and investigator are masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Onlay Mesh Reinforcement group (Active Comparator): The midline fascia was closed with running, slowly absorbable sutures (PDS 1-0) with a recommended suture length to wound length ratio of 4:1. An anterior plane with a width of about 8 cm was created between the anterior fascia and the subcutis. A Lightweight polypropylene mesh was used and placed on the anterior rectus fascia with an overlap of 3 cm. The mesh was fitted in the dissected space and it was fixed with PDS 2-0 suture. Fixing points are placed taking the mesh and the anterior fascia of the rectus muscle, at a distance of 3 cm between each point until completing its circunference.
  Interventions: Procedure: Mesh reinforcement
- RTL reinforcement group (Experimental): The RTL suture is placed parallel at a distance of 0.5 cm from the fascial margin. Ideally the thread should lie between the anterior and the posterior rectus muscle sheath; there should be no contact with the rectus muscle. A nonabsorbable monofilamental polypropylene thread and a 65-mm ½ needle are used. Around this longitudinal thread, the continuous suture for fascial closure is introduced immediately lateral to the thread; with running, slowly absorbable sutures (PDS 1-0) with a recommended suture length to wound length ratio of 4:1. An anterior plane with a width of about 8 cm was created between the anterior fascia and the subcutis
  Interventions: Procedure: RTL reinforcement

INTERVENTIONS:
Procedure: Mesh reinforcement — Once the surgery is over. The closure is made with the 4: 1 rule, then an onlay mesh is placed that exceeds 3 cm on each side the wound is fixed with suture.
  Other Names: Prophylactic Mesh reinforcement
  Arms: Onlay Mesh Reinforcement group
Procedure: RTL reinforcement — Once the surgery is finished, the ared is reinforced by placing a longitudinal suture parallel to the edge of the wound 0.5 cm, then the wound is closed with a 4: 1 rule but the suture enters lateral to the reinforcement suture
  Other Names: Technique RTL
  Arms: RTL reinforcement group

SUMMARY:
Introduction:

By definition, the laparotomy is a surgical incision into the abdomen cavity performed to examine the abdominal and retroperitoneal organs. The evisceration/eventration and the hernia are considered the most frequent complication of the midline laparotomy with a high morbidity and mortality related. Conditions that will require a second intervention, in Mexico represent the seventh cause of elective surgery and fourth cause of emergency procedures. The objective of this study is to determine if the incidence of post-incisional hernia in patients with high risk after a midline laparotomy are similar between the closure of the abdominal wall with the RTL technique and the supraaponeurotic mesh closure reinforcement.

Material and Methods: Clinical trial comparing the use of mesh against the RTL technique for post-incisional hernia prophylaxis. Two groups, triple blind Analysis will be carried out with intent to treat and not inferiority with 95% confidence intervals

DETAILED DESCRIPTION:
Introduction:

By definition, the laparotomy is a surgical incision into the abdomen cavity performed to examine the abdominal and retroperitoneal organs.

It is classified according to the medical indication: exploratory, therapeutic, stagemaker, and recently added "damage-control" laparotomy.

There exists so many ways to access the abdominal cavity, usually in relation with the organ or structure to treat; being classified in midline laparotomy, paramedian, transversal, oblique, abdominal-thoracic, etc.

Either an emergency or scheduled procedure, the more usual and functional continues being the midline laparotomy, since it allows a broader and faster approach, with less bleeding and easily to extend if it becomes necessary.

Both the evisceration/eventration and the hernia are considered the most frequent complication of the midline laparotomy with a high morbidity and mortality related. Conditions that will require a second intervention, in Mexico represent the seventh cause of elective surgery and fourth cause of emergency procedures.

So far only the use of the mesh has proven useful in reducing this complication. The authors published in 2016 a clinical trial where it showed that the technique is safe and effective to reduce the presence of incisional hernia, however the use of the mesh brings with it problems such as cost, possibility and use in contaminated cavities and postoperative pain. Therefore, the use of the RTL technique as an alternative means to this will help to have one more option for the management of patients with a high risk of incisional hernia.

Problem Statement:

Does the RTL closing technique in the midline laparotomy has the same incident of herniation than the close with supraaponeurotic mesh in patient with elevated risk?

Justification The presence of postincisional hernia need to be considerate as a serious disease, insomuch as it carry on highs rates of morbimortality. The presence of this eventuality is among 0.4-1.2% in elective surgery and up to 30% in emergency procedures.

It is calculated in de U.S.A. an approximate of 1 million of reinterventions a year to correct this condition, with the respective monetary, time and suffering cost to the patient and the health system.

Given the seriousness, the ultimate global consensus has determinate three main axes to the surgical community to board:

* Identify the relevance of the problem
* Improve the theoretical knowledge and technical capacity in the closing of the abdominal wall
* Implement prophylactic measures in the patients, especially in those with elevated risk.

With the present study the authors aim to contribute to this global recommendations, comparing two closing techniques of the abdominal wall after a midline laparotomy in patients with elevated risk of herniation. Both techniques are proved safe and useful in other studies, with no comparison to date.

Demonstrate that the use of RTL technique has a similar incidence of herniation than the mesh, in an attempt to prevent postincisional hernias after a midline laparotomy, will bring to the surgical community a cheaper and practical alternative to the mesh.

Objectives:

General:

To determinate if the incidence of post-incisional hernia in patients with high risk after a midline laparotomy are similar between the closure of the abdominal wall with the RTL technique and the supraaponeurotic mesh closure reinforcement.

Specifics:

* To identify the patients with high risk using de validated HERNIA-Project Score.
* To determinate the incidence of post-incisional hernia after one year of the initial midline laparotomy.
* To compare the incidence of post-incisional hernia between the two groups.
* To describe the complications related to each closure technique.

Hypothesis:

Ho Hypothesis:

There is no difference in the incidence of post-incisional hernia between the RTL technique and the reinforcement with supraaponeurotic mesh closure wall.

H1 Hypothesis:

There is difference in the incidence of post-incisional hernia between the RTL technique and the reinforcement with supraaponeurotic mesh closure wall.

Sample size:

The sample size was calculated according to the formula published by Bouemn et all 2015, and based on the results of Kholer and collaborators 2019, where the authors found in which a percentage of success was estimated with the standard treatment of 7% compared to the experimental management of 11%, with a margin of no less than 5%, with an alpha for a tail of 0.05%, and a beta of 20 %, a total of 125 patients per group was obtained.

Statistical analysis:

Categorical values will be present as frequency and percentage, comparisons between groups will be done using the χ2 test for binary data or Fisher´s exact test. Continuous variables will be presented as means (SDs) or median and range interquartile range, if they meet normal criteria and will be compared using the Mann-Whitney U-test or t student test. p-Values of less than 0.05 will be considered significant. Statistical analyses will be performed using SPSS statistical software, version 25.0.0 (IBM corp). Analysis by intention to treat will be used. A Kaplan-Meier curve of the occurrence of incisional hernias stratified by treatment group will be plotted, and a long-rank test will be used to compare the hernia incidence between the groups

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years undergoing midline laparotomy, independently of diagnostic or condition, elective or emergency surgery
* Patients with a score equal or greater than 7 of the hernia score
* Patients who accept to participate and sign the informed consent

Exclusion Criteria:

* Patients managed with open abdomen or with the impossibility of close the wall
* Patients who had a previous incisional hernia or patients who are participing in anohter trial
* Patients with a life expectative less than 12 months
* Pregnant patients Patients with the antecedent of rejection of prosthesic material

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with acute incisional hernia | 30 days
  An abdominal wall gap with or without bulge in the area of the postoperative scar palpable bi clinical examination (yes or not)
Number of participants with Incisional hernia | 1 year
  An abdominal wall gap with or without bulge in the area of the postoperative scar palpable bi clinical examination (yes or not)
Number of participants with Incisional hernia | 3 years
  An abdominal wall gap with or without bulge in the area of the postoperative scar palpable bi clinical examination (yes or not)

SECONDARY OUTCOMES:
Number of participants with surgical site infection | 30 days
  Includes at least one of the following: (a) purulent drainage is present (culture documentation not required); (b) organisms are isolated from fluid/tissue of the superficial incision; (c) at least one sign of inflammation (eg, pain or tenderness, induration, erythema, local warmth of the wound) is present; (d) the wound is deliberately opened by the surgeon; (e) the surgeon or clinician declares the wound infected
abdominal pain postoperative | 5 days postoperative
  It will be measured according to the visual analogue scale. Scale whose score goes from 0-10 being ten the maximum level expressed by the patient.
Number of participants with seroma | 10 days
  presence of accumulation of clear body fluids in a place where the tissue has been removed by surgery, not associated with infection

CONTACTS AND LOCATIONS:
Overall Officials: Jose de Jesus Alvarez Canales, Dr, Study Director — Hospital Regional de Alta Especialidad del Bajio
Locations (1):
- Hospital regional de Alta Especialidad del bajio, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Database available for analysis
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: previous sending of email requesting it

REFERENCES:
- [Background] Medina Ramírez O, Martínez Munive A. Hernias recurrentes y eventración posoperatoria. En: Consejo Mexicano de Cirugía General. Tratado de Cirugía General. Editorial Manual Moderno. México DF. 2009. p. 263-288
- [Background] Pelissier E, Armstrong O, Ngo P. Anatomía quirúrgica y vías de acceso del abdomen. EMC Elsevier Masson, Paris. 2011; 40-040: 1-40.
- [Background] Shell DH 4th, de la Torre J, Andrades P, Vasconez LO. Open repair of ventral incisional hernias. Surg Clin North Am. 2008 Feb;88(1):61-83, viii. doi: 10.1016/j.suc.2007.10.008. PMID 18267162
- [Background] van't RM, De Vos Van Steenwijk PJ, Bonjer HJ, Steyerberg EW, Jeekel J. Incisional hernia after repair of wound dehiscence: incidence and risk factors. Am Surg. 2004 Apr;70(4):281-6. PMID 15098775
- [Background] Ramirez Barba EJ, Lozano R, Lara Lona E. Epidemiologia de las hernias de la pared abdominal. En: Mayagoitia González JC, hernias de la pared abdominal. Tratamiento actual. 2 ed. Mexico; Editorial Alfil; 2009. p 9-11.
- [Background] Halm JA, Lip H, Schmitz PI, Jeekel J. Incisional hernia after upper abdominal surgery: a randomised controlled trial of midline versus transverse incision. Hernia. 2009 Jun;13(3):275-80. doi: 10.1007/s10029-008-0469-7. Epub 2009 Mar 4. PMID 19259615
- [Background] Le Huu Nho R, Mege D, Ouaissi M, Sielezneff I, Sastre B. Incidence and prevention of ventral incisional hernia. J Visc Surg. 2012 Oct;149(5 Suppl):e3-14. doi: 10.1016/j.jviscsurg.2012.05.004. Epub 2012 Nov 9. PMID 23142402
- [Background] Webster C, Neumayer L, Smout R, Horn S, Daley J, Henderson W, Khuri S; National Veterans Affairs Surgical Quality Improvement Program. Prognostic models of abdominal wound dehiscence after laparotomy. J Surg Res. 2003 Feb;109(2):130-7. doi: 10.1016/s0022-4804(02)00097-5. PMID 12643854
- [Background] van Ramshorst GH, Nieuwenhuizen J, Hop WC, Arends P, Boom J, Jeekel J, Lange JF. Abdominal wound dehiscence in adults: development and validation of a risk model. World J Surg. 2010 Jan;34(1):20-7. doi: 10.1007/s00268-009-0277-y. PMID 19898894
- [Background] Gómez CJ, Pere RC. Validación de un modelo de evisceración. Cir Esp. 2013. http://dx.doi.org/10.1016/j.ciresp.2012.12.0088
- [Background] Goodenough CJ, Ko TC, Kao LS, Nguyen MT, Holihan JL, Alawadi Z, Nguyen DH, Flores JR, Arita NT, Roth JS, Liang MK. Development and validation of a risk stratification score for ventral incisional hernia after abdominal surgery: hernia expectation rates in intra-abdominal surgery (the HERNIA Project). J Am Coll Surg. 2015 Apr;220(4):405-13. doi: 10.1016/j.jamcollsurg.2014.12.027. Epub 2015 Jan 2. PMID 25690673
- [Background] Cherla DV, Moses ML, Mueck KM, Hannon C, Ko TC, Kao LS, Liang MK. External Validation of the HERNIAscore: An Observational Study. J Am Coll Surg. 2017 Sep;225(3):428-434. doi: 10.1016/j.jamcollsurg.2017.05.010. Epub 2017 May 26. PMID 28554782
- [Background] Marwah S, Marwah N, Singh M, Kapoor A, Karwasra RK. Addition of rectus sheath relaxation incisions to emergency midline laparotomy for peritonitis to prevent fascial dehiscence. World J Surg. 2005 Feb;29(2):235-9. doi: 10.1007/s00268-004-7538-6. PMID 15654663
- [Background] Niggebrugge AH, Trimbos JB, Hermans J, Steup WH, Van De Velde CJ. Influence of abdominal-wound closure technique on complications after surgery: a randomised study. Lancet. 1999 May 8;353(9164):1563-7. doi: 10.1016/S0140-6736(98)10181-2. PMID 10334254
- [Background] Abbott DE, Dumanian GA, Halverson AL. Management of laparotomy wound dehiscence. Am Surg. 2007 Dec;73(12):1224-7. PMID 18186376
- [Background] Hollinsky C, Sandberg S. A biomechanical study of the reinforced tension line. A technique for abdominal wall closure and incisional hernias. European surgery. 2007. 39. 2. 122-127
- [Background] Hollinsky C, Sandberg S. Measurement of the tensile strength of the ventral abdominal wall in comparison with scar tissue. Clin Biomech (Bristol). 2007 Jan;22(1):88-92. doi: 10.1016/j.clinbiomech.2006.06.002. Epub 2006 Aug 10. PMID 16904247
- [Background] Hollinsky C, Sandberg S, Kocijan R. Preliminary results with the reinforced tension line: a new technique for patients with ventral abdominal wall hernias. Am J Surg. 2007 Aug;194(2):234-9. doi: 10.1016/j.amjsurg.2006.09.045. PMID 17618812
- [Background] Lozada-Hernandez EE, Mayagoitia-Gonzalez JC, Smolinski KR, AlvarezCanales JJ, Montiel Hinojosa L, Hernandez Villegas L. Comparacion de dos tecnicas de sutura para cierre aponeurotico en laparotomia media en pacientes con alto riesgo para evisceracion posquirurgica. Rev Hispanoamericana Hernia.2016; 4(4): 137-143
- [Background] Bhangu A, Fitzgerald JE, Singh P, Battersby N, Marriott P, Pinkney T. Systematic review and meta-analysis of prophylactic mesh placement for prevention of incisional hernia following midline laparotomy. Hernia. 2013 Aug;17(4):445-55. doi: 10.1007/s10029-013-1119-2. Epub 2013 May 28. PMID 23712289
- [Background] Lopez-Cano M, Pereira JA, Lozoya R, Feliu X, Villalobos R, Navarro S, Arbos MA, Armengol-Carrasco M. PREBIOUS trial: a multicenter randomized controlled trial of PREventive midline laparotomy closure with a BIOabsorbable mesh for the prevention of incisional hernia: rationale and design. Contemp Clin Trials. 2014 Nov;39(2):335-41. doi: 10.1016/j.cct.2014.10.009. Epub 2014 Nov 1. PMID 25445313
- [Background] Caro-Tarrago A, Olona Casas C, Jimenez Salido A, Duque Guilera E, Moreno Fernandez F, Vicente Guillen V. Prevention of incisional hernia in midline laparotomy with an onlay mesh: a randomized clinical trial. World J Surg. 2014 Sep;38(9):2223-30. doi: 10.1007/s00268-014-2510-6. PMID 24663481
- [Background] Jairam AP, Timmermans L, Eker HH, Pierik REGJM, van Klaveren D, Steyerberg EW, Timman R, van der Ham AC, Dawson I, Charbon JA, Schuhmacher C, Mihaljevic A, Izbicki JR, Fikatas P, Knebel P, Fortelny RH, Kleinrensink GJ, Lange JF, Jeekel HJ; PRIMA Trialist Group. Prevention of incisional hernia with prophylactic onlay and sublay mesh reinforcement versus primary suture only in midline laparotomies (PRIMA): 2-year follow-up of a multicentre, double-blind, randomised controlled trial. Lancet. 2017 Aug 5;390(10094):567-576. doi: 10.1016/S0140-6736(17)31332-6. Epub 2017 Jun 20. PMID 28641875
- [Background] Bouman AC, ten Cate-Hoek AJ, Ramaekers BL, Joore MA. Sample Size Estimation for Non-Inferiority Trials: Frequentist Approach versus Decision Theory Approach. PLoS One. 2015 Jun 15;10(6):e0130531. doi: 10.1371/journal.pone.0130531. eCollection 2015. PMID 26076354
- [Derived] Lozada Hernandez EE, Flores Gonzalez E, Chavarria Chavira JL, Hernandez Herrera B, Rojas Benitez CG, Garcia Bravo LM, Sanchez Rosado RR, Reynoso Gonzalez R, Gutierrez Neri Perez M, Reynoso Barroso MF, Soria Rangel J. The MESH-RTL Project for prevention of abdominal wound dehiscence (AWD) in high-risk patients: noninferiority, randomized controlled trial. Surg Endosc. 2024 Dec;38(12):7634-7646. doi: 10.1007/s00464-024-11358-w. Epub 2024 Oct 25. PMID 39453454

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT04134455/Prot_SAP_000.pdf